CLINICAL TRIAL: NCT01535313
Title: a Prospective Randomized Controlled Trial Comparing a Powered Bone Marrow Biopsy Device With a Manual System
Brief Title: Comparison of a Powered Bone Marrow Biopsy Device With a Manual System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Biopsycontrol
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Bone Marrow Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual (Hospital Systems TRAP Needle) (Active Comparator): Bone marrow biopsy with a standard manual system
  Interventions: Device: OnControl BM-Biopsy system
- Powered (Experimental)
  Interventions: Device: OnControl BM-Biopsy system

INTERVENTIONS:
Device: OnControl BM-Biopsy system — Bone marrow biopsy at posterior iliac crest
  Other Names: http://www.vidacare.com/OnControl/Bone-Marrow-Clinicians.aspx; http://www.hsmedicalinc.com/

SUMMARY:
Bone marrow biopsy quality as quantified by biopsy cylinder length and diagnostic usefulness is improved with a powered bone marrow biopsy device in comparison with a manual device.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* >= one previous bone marrow procedure
* INR > 1.4
* tThrombocyte count > 10 x109/l
* informed consent signed

Exclusion Criteria:

* cognitive impairment
* excessive tissue at anatomical landmarks
* BMI > 35 kg/m2
* allergy to premedication
* unable to lay flat in prone position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic usefulness (yes/no) of biopsy cylinder | within 1 week of biopsy
  The bone marrow biopsy cylinder is assessed by a pathologist who rates either "diagnostic" or "non diagnostic"

SECONDARY OUTCOMES:
patient pain during procedure | day 1 (two time points) and day 3-5
  patients underdoing biopsy rate the pain during, 15 min after and 3-5 days after the proceedure

CONTACTS AND LOCATIONS:
Overall Officials: Christoph M Bucher, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland